CLINICAL TRIAL: NCT05798780
Title: The ENHANCE Study: Exercise and Nutrition in Head And Neck CancEr Survivors: A Randomized Clinical Trial
Brief Title: The ENHANCE Study: Exercise and Nutrition in Head And Neck CancEr Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22330
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Oral Cavity Cancer; Oropharynx Cancer; Hypopharynx Cancer; Larynx Cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ENHANCE Intervention Diet and Excerise (Experimental): Participants will participate in 2 in-person supervised resistance training sessions every week for the 7 weeks (during radiation), followed by 2 ZOOM video conference supervised resistance training sessions every week for 5 weeks (after radiation). During radiation, participants will be provided 15 meals each week for 7 weeks. Participants will also attend weekly dietary coaching sessions. Participants will receive a Fitbit to wear continuously 24/7 over 12-weeks to track steps and activity intensity.
  Interventions: Behavioral: ENHANCE Intervention - Exercise and Nutrition
- ENHANCE Intervention Diet Only (Experimental): Participants will be provided 15 meals each week for 7 weeks that will accommodate common NIS concerns (ex. dysphagia and difficulty chewing) following an aMED dietary pattern (5 breakfast, 5 lunch, and 5 dinner), will be taught proper portion size, and will be asked to record percentages of each meal consumed in a provided food journal, in addition to any outside meals, snacks, or nutritional supplements. They will be provided with dietary coaching weekly to discuss NIS, aMED diet compliance, and set weekly SMART goals. Following completion of chemoradiotherapy (5 weeks), participants will be provided dietary coaching weekly (in-person or via videoconference), discuss NIS, aMED diet compliance at home, and set weekly SMART goals (30 min). Participants will receive a Fitbit to wear continuously 24/7 over 12-weeks to track steps and activity intensity.
  Interventions: Behavioral: ENHANCE Intervention - Nutrition Only
- Usual Care + Fitbit (No Intervention): Participants will receive handouts with diet and exercise education. Participants will receive a Fitbit to wear continuously 24/7 over 12-weeks to track steps and activity intensity.

INTERVENTIONS:
Behavioral: ENHANCE Intervention - Exercise and Nutrition — During radiation, participants will attend in-person supervised resistance training sessions once a week for 7 weeks, followed by 2 ZOOM video conference supervised resistance training sessions every week for 5 weeks, after radiation. Sessions will last approximately 30 minutes. During radiation, participants will be provided 15 meals each week for 7 weeks, 105 meals total. Participants will be asked to participate in 1 weekly dietary coaching session (in-person during radiation and video conference following radiation), create weekly SMART goals, follow an alternative Mediterranean diet pattern, and log all meals, snacks, and supplements consumed for the 12-week intervention.
  Arms: ENHANCE Intervention Diet and Excerise
Behavioral: ENHANCE Intervention - Nutrition Only — During chemoradiotherapy, participants will be provided 15 meals each week for 7 weeks (105 meals total) that will accommodate common NIS concerns (ex. dysphagia and difficulty chewing) following an aMED dietary pattern (5 breakfast, 5 lunch, and 5 dinner), will be taught proper portion size, and will be asked to record percentages of each meal consumed in a provided food journal, in addition to any outside meals, snacks, or nutritional supplements. They will be provided with dietary coaching weekly to discuss NIS, aMED diet compliance, and set weekly SMART goals (approximately 30 min). Following completion of chemoradiotherapy (5 weeks), participants will be provided dietary coaching weekly (in-person or via videoconference), discuss NIS, aMED diet compliance at home, and set weekly SMART goals (30 min). Trainers will monitor participants' Fitbit active minutes in real time throughout the intervention period and provide aerobic exercise encouragement accordingly.
  Arms: ENHANCE Intervention Diet Only

SUMMARY:
The purpose of the study is to design a physical activity and dietary intervention for head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Newly diagnosed tumors of the oral cavity, oropharynx, hypopharynx, or larynx
* No documented or observable psychiatric or neurological disorders that would interfere with study participation (e.g., dementia, psychosis)
* Able to speak and read English
* Able to consume food orally
* Willing to consume an alternative Mediterranean diet
* Scheduled to receive treatment with radiation or chemoradiation
* Screened via the Physical Activity Readiness Questionnaire (PAR-Q+) with medical clearance of treating physicians, as necessary
* Able to provide informed consent

Exclusion Criteria:

* Women who are pregnant
* Head and Neck Cancer not the primary diagnosis
* Patients scheduled to receive surgery
* Patients on enteral or parental nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Recruited - Feasibility | 12 Months
  The study will be deemed feasible if ≥ 60% of eligible participants are enrolled
Number of Participants who Complete Questionnaire - Retention - Feasibility | 12 weeks
  The study will be deemed feasible if ≥ 70% of participants complete post intervention questionnaire.
Participant Satisfaction of Timeline - Feasibility | 12 weeks
  The study will be deemed feasible if ≥ 70% of participants like the timing of the intervention using a likert scale (scale range Strongly agree to Strongly disagree)
Participant Average Attendance - Assessment Completion - Adherence | 12 weeks
  Participant assessment completion will be deemed successful if participant average attendance is ≥10 weeks of sessions (out of 12)
Number of Participants who Complete Task/Goals - Adherence | 12 weeks
  Study adherence will be deemed successful if ≥70% of participants report weekly tasks/goals adherence (e.g., gym and diet)
Participant Satisfaction Assessed with 5 Point Scale - Acceptability | 12 weeks
  Participants satisfaction will be measured using a 5 point scale (1 is the lowest, 5 is the highest) exit survey administered at the post-intervention follow-up.
Participant Intent to Continue Assessed with 5 Point Scale - Acceptability | 12 weeks
  Participants intent to continue will be measured using a 5 point scale (1 is the lowest, 5 is the highest) exit survey administered at the post-intervention follow-up.
Participant Knowledge Gained Assessed with 5 Point Scale - Acceptability | 12 weeks
  Participants knowledge gained will be measured using a 5 point scale (1 is the lowest, 5 is the highest) exit survey administered at the post-intervention follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Crowder, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=22330